CLINICAL TRIAL: NCT00041769
Title: A Phase II Randomized Controlled Trial Evaluating the Impact of Therapeutic Drug Monitoring (TDM) on Virologic Response to a Salvage Regimen in Subjects With a Normalized Inhibitory Quotient (NIQ) Less Than or Equal to 1 to One or More Protease Inhibitors
Brief Title: Using Drug Levels in the Blood to Guide Therapy in HIV Infected Patients Taking a Protease Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5146; AACTG A5146
Record Dates: First submitted 2002-07-16; First posted 2002-07-17 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2008-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Salvage Therapy; Viral Load; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Procedure: Therapeutic Drug Monitoring (TDM)

SUMMARY:
Drug resistance testing can be used to see which anti-HIV drugs are likely to suppress the growth of HIV and to select an anti-HIV regimen for HIV infected patients who have failed previous drug regimens. Therapeutic drug monitoring (TDM) is a process that involves measuring blood levels of a drug and may further increase the benefits that resistance testing offers by optimizing protease inhibitor (PI) drug concentrations. The purpose of this study is to determine whether changing the dose of PIs, as indicated by TDM, reduces the viral load in PI-experienced patients.

Hypothesis: Treatment-naive study participants who undergo TDM and whose clinicians' interpret their TDM results and adjust their PI doses will have better virologic response rates and decreased toxicities (and thus better treatment outcomes) than participants who do not undergo TDM.

DETAILED DESCRIPTION:
The use of drug resistance testing to guide the selection of an antiretroviral regimen for patients in whom current therapy is failing has gained growing acceptance in clinical practice. Genotypic and phenotypic resistance testing has been associated with improved short-term virologic outcome in prospective interventional trials. There is also growing evidence that monitoring drug levels, particularly of PIs, may add to the benefit provided by resistance testing. This study will assess the impact of TDM and resistance testing on lowering viral load in treatment-experienced patients and will also evaluate the mean change in plasma HIV RNA from study entry to Step 2 of the study.

No antiretrovirals will be provided by this study. Participants will be followed for a maximum of 48 weeks. Participants failing at least one combination antiretroviral regimen will have a screening drug resistance test performed while remaining on the failing regimen. In Step 1, participants will begin a salvage antiretroviral regimen within 7 days of study entry selected by their clinician using results of the resistance test. Two weeks after initiation of the salvage regimen, participants will have timed plasma samples obtained for PI trough levels. The results of the trough level tests will be used to calculate a normalized inhibitory quotient (NIQ) in order to determine eligibility for randomization into Step 2 at Week 4. Electrocardiograms (EKGs) and trough levels will be performed at Weeks 2, 6, and 10; support interviews to promote adherence will also be conducted by the study nurse or clinician at these times. Some participants taking tipranavir may have additional blood collection at Week 2.

In Step 2, participants with an NIQ of 1 or less will be randomly assigned to one of two arms. Arm A participants will receive standard care (SC) only, while participants in Arm B will receive SC plus dose-adjusted PIs based on the NIQ. Clinical and viral load assessment will be conducted at screening, entry, and Weeks 4, 10, 16, 24, 32, 40, and 48. Arm B participants will also have their PI trough levels checked at Weeks 6 and 10. Participants with an NIQ greater than 1 will be assigned to observational Arm C (open to up to 50 enrollees) or will stop their involvement in the study. Participants in Arms A, B, or C who have a viral load of 1000 copies/ml or higher or who experience virologic failure at or after Week 24 will be eligible to receive a second resistance test and enter Step 3.

Participants in Step 3 will begin a second salvage regimen; PI trough levels will be measured after 2, 6, and 10 weeks of salvage therapy. Those with an NIQ greater than 1, or with an NIQ of 1 or less and do not wish to escalate dose, will be followed on Step 3 for a maximum of 48 weeks after study entry.

All participants are encouraged to coenroll in ACTG A5128, Consent for Use of Stored Patient Specimens for Future Testing.

ELIGIBILITY:
Note: Enrollment into Arm C closed on 07/28/04 after reaching target accrual. Participants with a Week 2 NIQ of greater than 1 will be permanently discontinued from the study.

Inclusion Criteria for Step 1:

* HIV infected
* Viral load of 1000 copies/ml or more at study screening
* At least one viral load of 400 copies/ml or more within 6 months of study entry while on the failing antiretroviral regimen
* Virologic failure of at least one combination (two or more drugs) antiretroviral regimen, with at least one of these failing regimens containing a PI. Low dose ritonavir and hydroxyurea are not counted as antiretrovirals.
* Currently on a failing combination antiretroviral regimen
* Plan to initiate a salvage regimen containing a PI within 7 days of study entry
* Acceptable methods of contraception while receiving the study medications and for 6 weeks after stopping the medications. Participants who are currently taking efavirenz and who have undergone surgery to prevent conception (e.g., hysterectomy, tubal ligation, vasectomy) must provide physician's documentation of their current regimen and of their previous surgery.
* Resistance to at least one drug in the failing regimen, documented within 90 days of study entry
* Karnofsky performance scale of 70 or more within 30 days prior to study entry

Exclusion Criteria:

* Growth factors, interleukins, interferons (except for the treatment of hepatitis C), non-FDA approved systemic drugs, and HIV vaccines within 30 days of study entry
* Require certain medications prior to or during the study
* Certain heart conditions, if starting a PI-based regimen as the salvage regimen
* Acute illness or infection requiring treatment within 14 days of study entry
* Any condition that would limit ability to participate in the study
* Cancer requiring radiation or systemic chemotherapy
* Active drug or alcohol use or dependence that would interfere with the ability to meet study requirements
* Acute or chronic pancreatitis
* Planned use of hydroxyurea in the salvage regimen
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2002-06; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in log10 plasma HIV-1 RNA concentration from Step 2 entry (Week 4) to Week 24 (20 weeks post-randomization)
change in log10 plasma HIV-1 RNA concentration from study entry to Week 24 (20 weeks post-randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Demeter, MD, Study Chair — Infectious Diseases Unit, University of Rochester Medical Center; Mary Albrecht, MD, Study Chair — Division of Infectious Diseases, Beth Israel Deaconess Medical Center
Locations (47):
- United States (46):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Univ of California, San Diego Antiviral Research Center (AVRC), San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - San Mateo County AIDS Program, Stanford, California
  - Santa Clara Valley Med Ctr, Stanford, California
  - Willow Clinic, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Methodist Hosp of Indiana, Indianapolis, Indiana
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins Univ, Baltimore, Maryland
  - Harvard (Masschusetts General Hosp), Boston, Massachusetts
  - Beth Israel Deaconess-West Campus, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St. Louis Connect Care, St Louis, Missouri
  - Washington Univ (St. Louis), St Louis, Missouri
  - SUNY-Buffalo (Rochester), Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - Chelsea Clinic, New York, New York
  - New York University - Bellevue, New York, New York
  - Long Beach Memorial (Pediatric), New York, New York
  - Columbia Univ, New York, New York
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Ohio State Univ, Cincinnati, Ohio
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hosp, Providence, Rhode Island
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hosp, Providence, Rhode Island
  - Comprehensive Care Clinic, Nashville, Tennessee
  - Univ of Texas, Galveston, Galveston, Texas
  - Univ of Washington (Seattle), Seattle, Washington
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Clevenbergh P, Mouly S, Sellier P, Badsi E, Cervoni J, Vincent V, Trout H, Bergmann JF. Improving HIV infection management using antiretroviral plasma drug levels monitoring: a clinician's point of view. Curr HIV Res. 2004 Oct;2(4):309-21. doi: 10.2174/1570162043351129. PMID 15544452
- [Background] Duong M, Golzi A, Peytavin G, Piroth L, Froidure M, Grappin M, Buisson M, Kohli E, Chavanet P, Portier H. Usefulness of therapeutic drug monitoring of antiretrovirals in routine clinical practice. HIV Clin Trials. 2004 Jul-Aug;5(4):216-23. doi: 10.1310/NXJU-9ERQ-ADWW-UC5X. PMID 15472796
- [Background] Kiser JJ, Anderson PL, Gerber JG. Therapeutic drug monitoring: pharmacologic considerations for antiretroviral drugs. Curr HIV/AIDS Rep. 2005 Jun;2(2):61-7. doi: 10.1007/s11904-005-0020-8. PMID 16091250
- [Background] Rakhmanina NY, van den Anker JN, Soldin SJ. Therapeutic drug monitoring of antiretroviral therapy. AIDS Patient Care STDS. 2004 Jan;18(1):7-14. doi: 10.1089/108729104322740866. PMID 15006189
- [Background] Rendon A, Nunez M, Jimenez-Nacher I, Gonzalez de Requena D, Gonzalez-Lahoz J, Soriano V. Clinical benefit of interventions driven by therapeutic drug monitoring. HIV Med. 2005 Sep;6(5):360-5. doi: 10.1111/j.1468-1293.2005.00321.x. PMID 16156885
- [Result] DiFrancesco R, Rosenkranz S, Mukherjee AL, Demeter LM, Jiang H, DiCenzo R, Dykes C, Rinehart A, Albrecht M, Morse GD. Quality assessment for therapeutic drug monitoring in AIDS Clinical Trials Group (ACTG 5146): a multicenter clinical trial. Ther Drug Monit. 2010 Aug;32(4):458-66. doi: 10.1097/FTD.0b013e3181e4427a. PMID 20592644